CLINICAL TRIAL: NCT01171586
Title: mDiet: A Text Message Intervention for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA138730 (NIH)
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Overweight; Weight Loss
Keywords: Obesity; overweight; weight loss; weight maintenance; SMS; technology; cell phone; physical activity; nutrition
MeSH Terms: conditions — Overweight; Weight Loss; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SMS Only (Experimental): The SMS only group will receive hints, tips, strategies, and questions related to weight loss behaviors, physical activity, nutrition, and motivation. The messages will be "pushed" to participants (i.e. no response needed) and "pulled" from participants (i.e. response is needed). The SMS only group will also receive a brief printed or web based outline on weight loss resources and information.
  Interventions: Behavioral: mDiet
- SMS + Phone Counseling (Experimental): This group will receive hints, tips, strategies, and questions related to weight loss behaviors, physical activity, nutrition, and motivation. The messages will be "pushed" to participants (i.e. no response needed) and "pulled" from participants (i.e. response is needed). The group will also receive monthly counseling calls from a Health Coach to discuss barriers and solutions and will receive a brief printed or web based outline on weight loss resources and information.
  Interventions: Behavioral: mDiet
- Control (No Intervention): The Control group will receive a binder with an attractive set of Standard Print Materials related to weight loss that is comparable to what one would receive from community resources such as libraries, magazines and national non-profit or governmental organizations such as 5-A Day, American Heart Association and the like.

INTERVENTIONS:
Behavioral: mDiet — The goals of the intervention groups (SMS-only and SMS plus phone counseling) include: 5% weight loss, 500 k/cal per day deficit through reduced caloric intake and increased energy expenditure, 12,00 steps through the use of a pedometer, and a reduction in sedentary behaviors. Participants will receive daily "pushed" and "pulled" text messages, self-monitoring tools, and brief health promotion printed or wed materials on physical activity, nutrition, or other weight loss related topics.
  Arms: SMS + Phone Counseling; SMS Only

SUMMARY:
The purpose of the National Cancer Institute (NCI) funded randomized controlled study is to develop and evaluate a text message (SMS) based weight loss intervention to 309 overweight or moderately obese English and Spanish speaking adults ages 21 - 60. The investigators propose that participants randomized to the intervention arms will lose significantly more weight than those participants randomized to the control group.

DETAILED DESCRIPTION:
The SMS based intervention will be developed through formative research including focus groups, cognitive interviews, and a pilot test of a Spanish version of mDIET. The focus groups will be conducted with both English and Spanish speaking men and women to 1) learn more about the content areas to be addressed in the intervention including physical activity and sedentary behaviors to expand on previous research; 2) learn more about assessing equivalence and compatibility in intervention messages in English and Spanish; 3) identify the most culturally and linguistically appropriate messages; 4) assess text message use; 5) identify factors that influence food and physical activity decisions; and 6) identify health messages that Latinos see as most understandable, credible, and persuasive, cognitive interviews, and a pilot test of a Spanish version of mDIET. The cognitive interviews will be conducted in Spanish and will help inform translation of study materials (text messages and measures) from English to Spanish. An 8-week pilot test of the Latino (Spanish language) mDIET will be conducted to ensure that the text messages and SMS system works as expected in terms of usability and acceptability.

The randomized controlled trial will be a 12-month intervention with 309 study participants. Participants will be randomized to one of three groups: SMS-only, SMS plus phone counseling, and a control group (Details of the study arms are discussed in another section). The goals of the intervention groups (SMS-only and SMS plus phone counseling) include: 5% weight loss, 500 k/cal per day deficit through reduced caloric intake and increased energy expenditure, 12,00 steps through the use of a pedometer, and a reduction in sedentary behaviors. Participants will receive daily text messages, self-monitoring tools, and brief health promotion printed or wed materials on physical activity, nutrition, or other weight loss related topics. Participants will complete physiological and survey measures at baseline, 6 months, and 12 months to assess weight (BMI), physical activity and diet behaviors, psychosocial behaviors, environmental factors, and exposure and satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* Are 21 - 60 years
* Are overweight or moderately obese with a BMI between 27.0 - 39.9
* Have a cell phone that is capable of sending and receiving text and picture messages
* Have a permanent residence in San Diego County and intend to stay over the entire study duration
* Speak and read English or Spanish
* Are willing to attend all (3) measurement assessments at the research office
* Provide assent and have a legal guardian that will participate and provide parental permission/consent

Exclusion Criteria:

* Have any of the following conditions: pulmonary, cardiovascular, or musculoskeletal problems that would limit the ability to comply with moderate intensity physical activity (i.e. brisk walking)
* Are pregnant or intend to become pregnant during the study period
* Have a history of substance abuse
* Have a psychiatric disorder that would impair compliance with the study protocol
* Are using weight loss medications or supplements
* Are currently involved in another weight loss study or program

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 318 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 months
  To evaluate differences from baseline in percent weight loss at 12 months. We hypothesize that, compared to the usual care Standard Print condition differences in weight loss will be significant in both the SMS only (SMS = short message service or text message) and SMS+Phone intervention groups.

SECONDARY OUTCOMES:
Intervention Effects | 12 months
  To assess the intervention effects on weight loss by study group, diet, physical activity and sedentary behaviors, quality of life, and depression
Weight Loss Between Intervention Arms | 12 months
  To assess differences in weight loss between the 2 intervention arms (SMS only and SMS plus phone counseling)
Intervention Satisfaction and Exposure | 12 months
  To assess the level of satisfaction and use of the intervention components (SMS, phone counseling)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- UCSD, Atkinson Hall, 3rd Floor, La Jolla, California, United States

REFERENCES:
- [Derived] Godino JG, Golaszewski NM, Norman GJ, Rock CL, Griswold WG, Arredondo E, Marshall S, Kolodziejczyk J, Dillon L, Raab F, Jain S, Crawford M, Merchant G, Patrick K. Text messaging and brief phone calls for weight loss in overweight and obese English- and Spanish-speaking adults: A 1-year, parallel-group, randomized controlled trial. PLoS Med. 2019 Sep 25;16(9):e1002917. doi: 10.1371/journal.pmed.1002917. eCollection 2019 Sep. PMID 31553725
- [Derived] Kolodziejczyk JK, Norman GJ, Roesch SC, Rock CL, Arredondo EM, Madanat H, Patrick K. Exploratory and confirmatory factor analyses and demographic correlate models of the strategies for weight management measure for overweight or obese adults. Am J Health Promot. 2015 Mar-Apr;29(4):e147-57. doi: 10.4278/ajhp.130731-QUAN-391. Epub 2014 Mar 26. PMID 24670075
- [Derived] Kolodziejczyk JK, Norman GJ, Barrera-Ng A, Dillon L, Marshall S, Arredondo E, Rock CL, Raab F, Griswold WG, Sullivan M, Patrick K. Feasibility and effectiveness of an automated bilingual text message intervention for weight loss: pilot study. JMIR Res Protoc. 2013 Nov 6;2(2):e48. doi: 10.2196/resprot.2789. PMID 24200517